CLINICAL TRIAL: NCT03808714
Title: Development, Implementation, and Evaluation of a Smoking Cessation Tailored to Rural Young Adult African American Men: Toward Scalability
Brief Title: Smoking Cessation Tailored to Rural Young Adult African American Men:
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruitment due to COVID-19
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Isabel Scarinci, Primary Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-160204003
Record Dates: First submitted 2019-01-16; First posted 2019-01-17 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Smoking Cessation
Keywords: african american, smoking cessation, rural, young adults
MeSH Terms: conditions — Smoking Cessation | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Intervention - smoking cessation program delivered by Community Health Worker with pharmacological support by a specialist at the university Control - Alabama Quitline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): We expect the intervention to consist of 3 to 4 group sessions and at least one individual session (delivered by a trained Community Health Worker) plus pharmacological consultation(s) via telemedicine, but this will be determined during pretesting.
  Interventions: Behavioral: TOUCHDOWN
- Control (Active Comparator): Alabama Tobacco Quitline, which is considered the "standard-of-care" for smoking cessation in Alabama.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: TOUCHDOWN — We expect the intervention to consist of 3 to 4 group sessions and at least one individual session plus pharmacological consultation(s) via Skype, but this will be determined during pretesting. CHWs will have IPads with cellular connectivity and will be present when the pharmacological approach is discussed with the participant so that they can reinforce the message with the participant and be the liaisons between the participant and physician.
  Arms: Intervention
Behavioral: Control Group — Alabama Quitline
  Arms: Control

SUMMARY:
Our preliminary data shows that 39.9% of AA men between 19 and 30 years of age who resided in rural Alabama smoke cigarettes. Although it has been well established that a combination of pharmacotherapy and advice-oriented counseling and/or cognitive behavioral interventions are efficacious in promoting smoking cessation across diverse populations, these evidence-based treatments for tobacco dependence have not proven to be effective/efficacious (or even accessible) among some subpopulations suffering disproportionally from tobacco-related morbidity and mortality. The overall goal of this feasibility study is to make adaptations to these evidence-based approaches, and develop, implement, and examine the feasibility and scalability of a theory-based, culturally relevant smoking cessation intervention for young adult AA men in rural Alabama who smoke cigarettes. Our formative assessments point to a cognitive-behavioral intervention delivered by a trained Community Health Worker with the support from an "expert" physician who can deliver the pharmacological component via Skype through an integrated approach. The proposed study will address the next three steps in this process: development of the intervention, pretesting, and feasibility. First, we will develop the intervention with input from a Community Advisory Committee, followed by an iterative process by which the target audience will be exposed to materials and messages to provide feedback (pretesting). Once all intervention components are finalized, we will recruit participants, randomly assign them to intervention/control groups, pilot test, and evaluate the intervention. The comparison group will be the Alabama Tobacco Quitline with 8 weeks of Nicotine Replacement Therapy to be consistent with the pharmacological approach proposed for the intervention. The primary outcome will be 7-day point prevalence abstinence (defined as no cigarettes in the past 7 days and verified through measurement of exhaled carbon monoxide levels) at 6-month follow-up. We will also conduct detailed treatment fidelity and scalability assessments (acceptability, feasibility, potential reach and adoption, alignment with the strategic context) to inform a full-scale efficacy trial.

DETAILED DESCRIPTION:
Despite smoking fewer cigarettes daily, African American (AA) men suffer higher morbidity and mortality associated with tobacco-related disorders than whites. Our preliminary data shows that 39.9% of AA men between 19 and 30 years of age who resided in rural Alabama smoke cigarettes. Although it has been well established that a combination of pharmacotherapy and advice-oriented counseling and/or cognitive behavioral interventions are efficacious in promoting smoking cessation across diverse populations, these evidence-based treatments for tobacco dependence have not proven to be effective/efficacious (or even accessible) among some subpopulations suffering disproportionally from tobacco-related morbidity and mortality. The overall goal of this feasibility study is to make adaptations to these evidence-based approaches, and develop, implement, and examine the feasibility and scalability of a theory-based, culturally relevant smoking cessation intervention for young adult AA men in rural Alabama who smoke cigarettes. Our formative assessments point to a cognitive-behavioral intervention delivered by a trained Community Health Worker with the support from an "expert" physician who can deliver the pharmacological component via Skype through an integrated approach. The proposed study will address the next three steps in this process: development of the intervention, pretesting, and feasibility. First, we will develop the intervention with input from a Community Advisory Committee, followed by an iterative process by which the target audience will be exposed to materials and messages to provide feedback (pretesting). Once all intervention components are finalized, we will recruit participants, randomly assign them to intervention/control groups, pilot test, and evaluate the intervention. The comparison group will be the Alabama Tobacco Quitline with 8 weeks of Nicotine Replacement Therapy to be consistent with the pharmacological approach proposed for the intervention. The primary outcome will be 7-day point prevalence abstinence (defined as no cigarettes in the past 7 days and verified through measurement of exhaled carbon monoxide levels) at 6-month follow-up. We will also conduct detailed treatment fidelity and scalability assessments (acceptability, feasibility, potential reach and adoption, alignment with the strategic context) to inform a full-scale efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

(a) African American; (b) men; (c) between the ages of 18 and 30; (d) residing in Sumter and Greene counties; and (e) smoked cigarettes within the past seven days. For the feasibility testing of the intervention, participants must have a permanent residence in the county and no intent to move within the next 12 months.

Exclusion Criteria:

* Recent MI and unstable angina.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — African American men between the ages of 18 and 30 living in the participating rural counties
Enrollment: 35 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Cessation | 6 months
  The primary outcome will be a 7-day point prevalence abstinence (defined as no cigarettes in the past 7 days and verified through measurement of exhaled carbon monoxide levels) at 6-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel C Scarinci, PhD, Principal Investigator — University of Alabama at Birmingham; William Carroll, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No